CLINICAL TRIAL: NCT00875095
Title: Impact of Sperm DNA Integrity on ART Treatment
Brief Title: Impact of Sperm DNA Integrity on Artificial Reproductive Treatment (ART)
Status: Terminated | Type: Observational
Why Stopped: Study funding was withdrawn by the sponsor following agreement that slow patient recruitment warranted a new approach.
Sponsor: Northwell Health (Other)
Collaborators: Organon (Industry)
Responsible Party: Principal Investigator, Dennis Marchesi, laboratory supervisor, Northwell Health
Other Study IDs: 07.08.118
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Sperm DNA Impact on ART Outcomes
Keywords: sperm DNA integrity; Toluidine blue staining

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Smears of semen samples will be stained and stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IUI patients: Patients undergoing routine semen analysis as part of their infertility treatment pertaining to success or failure with intrauterine insemination, based upon their sperm DNA integrity
- IVF patients: Couples undergoing routine screening prior to IVF retrievals to assess their reproductive treatment outcomes as compared to the sperm DNA integrity

SUMMARY:
The purpose of this study is to establish a new criteria with which to judge the quality of sperm samples submitted for artificial reproductive treatments. It is believed that this type of testing can compliment the traditional semen analysis to better drive patient care.

ELIGIBILITY:
Inclusion Criteria:

* needs interventions through artificial reproductive treatment to achieve a pregnancy

Exclusion Criteria:

* severly oligozoospermic patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient population at the Center for Human Reproduction.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Sperm DNA integrity | 1 day

SECONDARY OUTCOMES:
achievement of a successful pregnancy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Avner Hershlag, MD, Principal Investigator — Northwell Health; Dennis E Marchesi, MSc, Study Director — Northwell Health
Locations (1):
- The Center for Human Reproduction, Manhasset, New York, United States

REFERENCES:
- [Background] Andreetta AM, Stockert JC, Barrera C. A simple method to detect sperm chromatin abnormalities: cytochemical mechanism and possible value in predicting semen quality in assisted reproductive procedures. Int J Androl. 1995 Jun;18 Suppl 1:23-8. doi: 10.1111/j.1365-2605.1995.tb00634.x. PMID 7558384
- [Background] Chohan KR, Griffin JT, Lafromboise M, De Jonge CJ, Carrell DT. Comparison of chromatin assays for DNA fragmentation evaluation in human sperm. J Androl. 2006 Jan-Feb;27(1):53-9. doi: 10.2164/jandrol.05068. PMID 16400078
- [Background] Erenpreiss J, Jepson K, Giwercman A, Tsarev I, Erenpreisa J, Spano M. Toluidine blue cytometry test for sperm DNA conformation: comparison with the flow cytometric sperm chromatin structure and TUNEL assays. Hum Reprod. 2004 Oct;19(10):2277-82. doi: 10.1093/humrep/deh417. Epub 2004 Jul 22. PMID 15271869
- [Background] Erenpreisa J, Erenpreiss J, Freivalds T, Slaidina M, Krampe R, Butikova J, Ivanov A, Pjanova D. Toluidine blue test for sperm DNA integrity and elaboration of image cytometry algorithm. Cytometry A. 2003 Mar;52(1):19-27. doi: 10.1002/cyto.a.10015. PMID 12596248
- [Background] Erenpreiss J, Bars J, Lipatnikova V, Erenpreisa J, Zalkalns J. Comparative study of cytochemical tests for sperm chromatin integrity. J Androl. 2001 Jan-Feb;22(1):45-53. PMID 11191087
- [Background] Gavrieli Y, Sherman Y, Ben-Sasson SA. Identification of programmed cell death in situ via specific labeling of nuclear DNA fragmentation. J Cell Biol. 1992 Nov;119(3):493-501. doi: 10.1083/jcb.119.3.493. PMID 1400587
- [Background] Said TM, Mahfouz R, Erenpreiss J, Giwercman A, Sharma RK, and Agarwal A. Association of intermediate staining patterns using the Toluidine blue test with late apoptosis and necrosis in human spermatozoa. 2006 Online ASRM abstract submission #06-A-1199-ASRM
- [Background] Said TM, Agarwal A, Erenpreiss J, Mahfouz R, Giwercman A, and Evenson DP. Evaluation of seminal fractions using Toluidine blue test and sperm chromatin structure assay. 2006 Online ASRM abstract submission #06-A-1123-ASRM
- [Background] Schlegel PN, Paduch DA. Yet another test of sperm chromatin structure. Fertil Steril. 2005 Oct;84(4):854-9. doi: 10.1016/j.fertnstert.2005.04.050. PMID 16213834
- [Background] World Health Organization (1999) WHO Laboratory manual for the examination of human semen ana sperm-cervical mucus interactions. 4rth ed. prepared by the WHO special programmed of research, development and research training in human reproduction. Cambridge University Press.